CLINICAL TRIAL: NCT06821633
Title: Investigating the Retardation Effect of OCTA-Guided Targeted Photocoagulation on the Progression of Non-Perfusion Areas in Diabetic Retinopathy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jie Li, Principal Investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-KY740-1
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eyes with NPDR that were diagnosed and underwent TRP guided by OCTA at our hospital (Experimental): The patient's eyes were first scanned using the Topcon OCTA (five-field montage) with a 24×20mm and a 6×6mm scan range. After enrollment, the patient underwent treatment on the same day in the retinal laser room. The laser treatment was performed by the same ophthalmologist. After obtaining baseline fundus images, the treating ophthalmologist overlaid the OCTA images onto the fundus images using retinal vessel alignment to guide targeted photocoagulation of the retinal non-perfusion (NP) areas under OCTA guidance. The specific photocoagulation method involved applying a grid pattern of spot laser (3×3) to the NP area once, with the treatment area extending beyond the NP boundary by one laser spot diameter. The total procedure duration was 10-20 minutes.
  Interventions: Procedure: Targeted laser photocoagulation guided by OCTA (Optical Coherence Tomography Angiography)
- Eyes with NPDR that were diagnosed at our hospital (No Intervention): Perform the same examination but administer no treatment

INTERVENTIONS:
Procedure: Targeted laser photocoagulation guided by OCTA (Optical Coherence Tomography Angiography) — The patient's eyes were first scanned using the Topcon OCTA (five-field montage) with a 24×20mm and a 6×6mm scan range. After enrollment, the patient underwent treatment on the same day in the retinal laser room. The laser treatment was performed by the same ophthalmologist. After obtaining baseline fundus images, the treating ophthalmologist overlaid the OCTA images onto the fundus images using retinal vessel alignment to guide targeted photocoagulation of the retinal non-perfusion (NP) areas under OCTA guidance. The specific photocoagulation method involved applying a grid pattern of spot laser (3×3) to the NP area once, with the treatment area extending beyond the NP boundary by one laser spot diameter. The total procedure duration was 10-20 minutes.
  Arms: Eyes with NPDR that were diagnosed and underwent TRP guided by OCTA at our hospital

SUMMARY:
This study aims to evaluate the impact of widefield OCTA-guided selective photocoagulation on the progression of diabetic retinopathy (DR) by comparing the control of non-perfusion (NP) areas, DR grading, and management of other DR lesions. The study is designed as a parallel randomized controlled trial. From February 2025 to August 2026, 30 diabetic patients attending the Ophthalmology Department of Sichuan Provincial People's Hospital will be enrolled. Using a simple randomization method, one eye of each patient will be assigned to the intervention group, while the contralateral eye will serve as the control, resulting in 30 eyes in each group. The intervention group will undergo OCTA-guided selective photocoagulation, specifically using a grid pattern (3x3) of spot laser applied once to the NP area, extending one spot diameter beyond the NP boundary. Each session will last 10-20 minutes. The control group will receive no treatment. The study will compare changes in NP area, DR grading progression, and control of other DR lesions at 3, 6, 9, and 12 months between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Type 1 or Type 2 diabetes mellitus
* Clinical dilated fundus examination and Optos imaging within 7 fields showing diabetic retinopathy (DR) lesions no more severe than severe non-proliferative diabetic retinopathy (NPDR)
* Optical coherence tomography angiography (OCTA) demonstrating non-perfusion (NP) areas greater than 1 disc diameter (PD) in both eyes
* Diabetic retinopathy in both eyes at the same stage, with the total NP area within the observed range of OCTA being comparable (difference less than 5 PD)
* Absence of other ocular diseases that could lead to the formation of retinal microaneurysms
* Absence of other ocular diseases that could lead to the formation of retinal non-perfusion areas
* No diabetic macular edema involving the fovea
* No history of retinal laser treatment
* No history of intravitreal injection therapy within the past 3 months
* No history of ocular surgery other than cataract surgery
* Ability to cooperate with all examinations and provide informed consent

Exclusion Criteria:

* Optical media opacity affecting OCTA imaging
* Patients with difficulties in cooperating with laser treatment
* Patients with renal failure, diabetic neuropathy, or severe cardiovascular diseases
* Patients who are unlikely to complete follow-ups every 3 months, as well as those residing in other provinces
* Patients requiring early PRP (conditions include: combined DME, planned cataract surgery, pregnancy planning, early PDR, poor follow-up compliance, severe vision loss in the other eye, poor glycemic control, poor renal function, or type 1 diabetes)
* FFA showing NP greater than 10 PD within the ETDRS area or a total NP area greater than 75 PD, or an ischemia index greater than 35%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2026-08-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
The area size of NP (in PD units) in two groups of eyes at 0, 3, 6, 9, and 12 months | From enrollment to reexamination at 0,3,6,9, and 12 months

SECONDARY OUTCOMES:
The number of microaneurysms, intraretinal microvascular abnormalities (IRMA) in both groups of eyes at 0, 3, 6, 9, and 12 months | From enrollment to reexamination at 0,3,6,9, and 12 months
The number of neovascularization (NV) in both groups of eyes at 0, 3, 6, 9, and 12 months | From enrollment to reexamination at 0,3,6,9, and 12 months
Area of foveal avascular zone (FAZ) at 0, 3, 6, 9, and 12 months in two groups of eyes | From enrollment to reexamination at 0,3,6,9, and 12 months
DR grading at 0, 3, 6, 9, and 12 months in two groups of eyes | From enrollment to reexamination at 0,3,6,9, and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
2030, via https://pan.baidu.com
Supporting Information: CSR
Time Frame: 2025 and forever
Access Criteria: via https://pan.baidu.com
URL: http://pan.baidu.com